CLINICAL TRIAL: NCT05051527
Title: Observational, Single Arm, Prospective Study to Evaluate the Effectiveness of Legalon® in Addition to Diet and Exercise in Reducing Plasma Levels of Liver Enzymes
Brief Title: Study to Evaluate the Effectiveness of Legalon®
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: Meda Pharma S.p.A. (Unknown)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: 2019-24-NIS-Multicountry-3327
Record Dates: First submitted 2021-09-07; First posted 2021-09-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Silymarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Legalon®: Legalon® 140 mg
  Interventions: Drug: Legalon® 140 mg

INTERVENTIONS:
Drug: Legalon® 140 mg — Legalon® 140 mg as per the Summary of Product Characteristics (SPC) and as per treating Investigator's decision

SUMMARY:
This is a multinational, multicentre, prospective, non-interventional study (NIS) in non-alcoholic fatty liver disease (NAFLD) patients with concomitant metabolic syndrome treated with Legalon® combined with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Legalon® monotherapy prescribed by the treating Investigator according to the SPC, independently from and within a 4-week window prior to enrolment into the study.
2. Male/female, 18 years of age and older
3. Able to provide informed consent
4. Available baseline blood results not older than 4 weeks from inclusion, with elevated plasma level of at least one liver enzyme with respect to normal ranges of local laboratory (>1 UNL)
5. NAFLD diagnosed by ultrasonography according to the protocol by Hamaguchi or by the protocol of Ballestri
6. Presence of metabolic syndrome, defined as the presence of at least 3 out of 5 of the following:

   1. Central obesity (for Asian population, waist circumference ≥90 cm in males, ≥80 cm in females)
   2. Insulin resistance (fasting blood glucose ≥100mg/dl or under medication)
   3. High blood pressure (≥ 130/85 mmHg or on medication)
   4. High triglycerides (≥150 mg/dl or on medication)
   5. Low HDL-cholesterol (<40mg/dl in men, <50mg/dl in women)
7. Started diet and exercise interventions, as per treating Investigator's suggestion and in line with current guidelines within a 4-week window prior to enrolment into the study

Exclusion Criteria:

1. Significant alcohol intake >7 standard alcoholic drinks per week (70 g ethanol) in women and >14 (140 g) in men
2. Received Legalon® or any other hepatoprotective treatment before the allowed 4-week window prior to enrolment into the study.
3. On diet and exercise before the allowed 4-week window prior to enrolment into the study.
4. Other concomitant established / diagnosed liver diseases, including chronic hepatitis B, chronic hepatitis C, autoimmune liver diseases (including autoimmune hepatitis), celiac disease, primary biliary cholangitis, primary sclerosing cholangitis, biliary obstruction, drug-induced liver disease (including herbal medicines and dietary supplements), metabolic liver disorders (such as Wilson's disease, alpha-1- antitrypsin deficiency, hemochromatosis, glycogen storage disorders, cholesterol storage disorders), severe liver diseases, non-alcoholic steatohepatitis (NASH) or other forms of advanced fatty liver disease (including clinically relevant fibrosis, >F2, or established cirrhosis), liver carcinoma
5. Patients treated with drugs with known hepatotoxic effects (at risk of drug-induced liver injury [DILI]), including herbal medicines and dietary supplements
6. Other major diseases that, in the treating Investigator opinion, can impair liver function, as for example type 1 diabetes
7. Pregnant and/or breastfeeding women
8. Persons that, in treating Investigator's opinion, are not able to fulfil study requirements
9. Persons that refuses to participate
10. Patients that, in the Investigator's opinion, are or have been infected with COVID-19 (i.e. presence/referral of COVID-19 symptoms or positive antigenic/molecular test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-alcoholic fatty liver disease and concomitant metabolic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of Legalon® | 6 months
  - To observe the effectiveness of Legalon® in addition to diet and exercise in lowering the plasma levels of liver enzymes in patients with non-alcoholic fatty liver disease (NAFLD) and concomitant metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Lee Yeong Yeh, Dr., Principal Investigator — Department of Medicine, Hospital Universiti Sains Malaysia,16150 Kelantan Darul Naim, MALAYSIA; Sakkarin Chirapongsathorn, Dr., Principal Investigator — Department of Internal Medicine, Phramongkutklao Hospital, Bangkok, 40002, Thailand; Marilyn Arguillas, Dr., Principal Investigator — Davao Doctors Hospital, Davao City, Philippines 8000
Locations (1):
- Phramongkutklao Hospital, 315 Ratchawithi Rd, Thung Phaya Thai, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No